CLINICAL TRIAL: NCT06718985
Title: Does Incorporating Bone Mineral Density Change Fracture Risk Assessment and Influence Treatment Decisions in Rheumatoid Arthritis Patients?
Brief Title: Impact of Bone Mineral Density on Fracture Risk Assessment in RA
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Fatma Nur Kesiktaş, Principle Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstPRMTRH55
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study investigates whether incorporating bone mineral density (BMD) into FRAX calculations changes fracture risk assessment and influences treatment decisions in rheumatoid arthritis (RA) patients. Analyzing 60 RA patients, FRAX scores for 10-year major osteoporotic and hip fractures were calculated with and without BMD. While no significant differences were found between the two methods, discrepancies in treatment recommendations were identified, particularly for hip fractures. The findings emphasize the importance of combining BMD and FRAX for a more comprehensive fracture risk assessment and informed treatment decision-making in RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) based on ACR/EULAR criteria.
* Age between 40-90 years.
* Dual-energy X-ray absorptiometry (DXA) results obtained within the past six months.
* Availability of complete clinical and demographic data for fracture risk assessment.
* Patients who provide informed consent for the study.

Exclusion Criteria:

* Patients with secondary causes of osteoporosis (e.g., hyperparathyroidism, Cushing's syndrome).
* Use of medications affecting bone metabolism (e.g., glucocorticoids >7.5 mg/day, bisphosphonates, denosumab) within the past year.
* History of metabolic bone diseases other than osteoporosis (e.g., osteomalacia, Paget's disease).
* Patients with a history of malignancy, except for non-melanoma skin cancer.
* Incomplete or missing data required for FRAX or DXA analysis.
* Any condition or comorbidity likely to affect fracture risk assessment, as determined by the clinician.

Ages: 40 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-12-04 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Concordance Between FRAX Scores With and Without BMD | 0 day
  The agreement between 10-year fracture risk calculations for major osteoporotic fractures (MOF) and hip fractures (HF) using FRAX with and without bone mineral density (BMD).

SECONDARY OUTCOMES:
Treatment Threshold Exceedance Based on FRAX Calculations | 0 day
  Proportion of patients exceeding treatment thresholds for MOF and HF risk based on FRAX calculations with and without BMD.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, Bahcelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No